CLINICAL TRIAL: NCT07113509
Title: Randomized Clinical Study for Printed Definitive Hybrid Resin Implant Crowns: Short-term Effects of Surface Finishing and Wear
Brief Title: Clinical Trial for Printed Implant Resin Crowns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Mine Dundar Comlekoglu, Prof. Dr., Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07.06.2022-No: 22-5.1/57
Record Dates: First submitted 2025-07-25; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Surface Finish; Wear
Keywords: glazing; mechanical polishing; printed implant hybrid resin crowns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mechanical polishing (Active Comparator): surface finishing with mechanical polishing
  Interventions: Procedure: mechanical polishing
- glazing (Active Comparator): glaze liquid application and curing
  Interventions: Procedure: glazing

INTERVENTIONS:
Procedure: mechanical polishing — mechanical polishing of implant resin crowns with polishing paste and discs
  Arms: mechanical polishing
Procedure: glazing — glaze liquid application followed by light-curing of the resin implant crowns
  Arms: glazing

SUMMARY:
The goal of this clinical trial is to assess the clinical performance of printed resinous implant crowns with two surface finishing protocols-mechanical polishing versus glazing. Qualitative performance will be checked by scoring systems.

The main questions it aims to answer are;

* Do printed resin implant crowns clinically succeed in the sort-term?
* Do mechanical polishing or glazing the crowns would be better for clinical performance?

Participants will:

* receive either mechanically polished or glazed printed resin implant crowns,
* visit at 6-months and 1 year for clinical check

DETAILED DESCRIPTION:
Wear amounts of the printed resin implant crowns will be measured

ELIGIBILITY:
Inclusion Criteria:

* single-tooth edentulism
* no head/neck radiotherapy or bisphosphonate/denosumab therapy
* adequate alveolar crest width (implant diameter + 3 mm)
* absence of active periodontal disease, and willingness to comply.

Exclusion Criteria:

* ASA class III
* heavy smoking (>20 cigarettes/day)
* pregnancy or lactation
* allergies to titanium
* need for hard or soft tissue augmentation
* bisphosphonate/denosumab therapy
* head/neck radiotherapy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
printed resin implant crown survival | From enrollment to the end of treatment at 6 months
  survival with repairable failures
no catastrophic failure of the printed resin implant crowns | 6 months
  clinical performance with repairable failures

CONTACTS AND LOCATIONS:
Overall Officials: Ercan Yigit, PhD, Principal Investigator — Ege University
Locations (1):
- Ege University Faculty of Dentistry, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: rationale and reference for the study set up — https://pubmed.ncbi.nlm.nih.gov/38541534/